CLINICAL TRIAL: NCT04785456
Title: Repetitive Transcranial Magnetic Stimulation for Suicidality in Opioid Use Disorders
Brief Title: rTMS for Suicidality in Opioid Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 131/2020
Record Dates: First submitted 2021-02-12; First posted 2021-03-08 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Major Depressive Disorder; Opioid-use Disorder
Keywords: Suicidality; rTMS
MeSH Terms: conditions — Depressive Disorder, Major; Opioid-Related Disorders; Suicidal Ideation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active TBS (Experimental): Daily, 4-week, 5-days per week treatment sessions, each consisting of:
  First, intermittent TBS (iTBS) over the L-DLPFC: triplet 50 Hz bursts, repeated at 5 Hz, 2 s on and 8 s off, (600 pulses per session, total duration of 3 min 9 s), then continuous TBS (cTBS) over the R-DLPFC as 40 s uninterrupted bursts (600 pulses). Intensity at 120% resting motor threshold (RMT).
  Interventions: Device: Active TBS
- Sham TBS (Sham Comparator): Daily, 4-week, 5-days per week treatment sessions. The sham coil will generate auditory and somatosensory (vibratory) stimuli identical to the active stimulation.
  Interventions: Device: Sham TBS

INTERVENTIONS:
Device: Active TBS — MagPro X100 device equipped with a Cool-B70 A/P coil and Qooler fluid-cooling device (MagVenture, Farum, Denmark)
  Arms: Active TBS
Device: Sham TBS — MagPro X100 device equipped with a Cool-B70 A/P coil and Qooler fluid-cooling device (MagVenture, Farum, Denmark)
  Arms: Sham TBS

SUMMARY:
This trial is a randomized, double blind, controlled pilot study that will compare bilateral theta burst stimulation (TBS) and sham treatment for patients with opioid use disorder (OUD) and Major Depressive Disorder (MDD) experiencing suicidality.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) to the dorsolateral prefrontal cortex (DLPFC) is used therapeutically in major depressive disorder resistant to standard treatments, and recently also shown to be effective in reducing suicidality with a bilateral approach. Recently, a new form of rTMS has been developed called theta burst stimulation (TBS) which requires a much shorter daily treatment duration and has been found to be non-inferior to standard rTMS. The investigators propose to conduct a randomized controlled clinical trial of a daily, 20 session course of bilateral TBS versus sham stimulation in the treatment of suicidality in patients with OUD and MDD. The investigators will explore whether TBS can have other clinical effects on decreasing symptoms of MDD, craving for opioids, and rates of relapse to opioid use. The investigators will also examine whether rTMS can engage GABA mediated inhibition using combined transcranial magnetic stimulation and electroencephalography (TMS-EEG) will be assessed before and after intervention. Clinical outcomes measured before, during, at end of treatment, and 4-weeks post treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of providing informed consent and research procedures according to the brain stimulation attending psychiatrist
2. Between the ages of 18-60 years
3. Mini-International Neuropsychiatric Interview (MINI) confirmed diagnosis of Opioid Dependence and MDD.
4. On a stable treatment regimen without any change in opioid agonist or antidepressant medications or dosages in the last 30 days. Participants will be asked not to change their medication regimen for the duration of the study.
5. Baseline score of >/=4 on the scale for suicidal ideation (SSI).

Exclusion Criteria:

1. Currently pregnant or intending to be pregnant during the duration of the study
2. Bipolar disorder, any psychotic disorder or current psychotic symptoms
3. Previous rTMS treatment
4. Known active seizure disorder, significant head injury with an imaging verified lesion
5. Unstable medical illness
6. Presence of cardiac pacemaker, intracranial implant, or metal in the cranium
7. Participants taking > 2 mg lorazepam (or a benzodiazepine at an equivalent dose) or taking any anticonvulsant medication during treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Scale for Suicidal Ideation Remission | Change from baseline, to end of TBS treatment course (4 weeks), and at 1 month follow up
  A semi-structured interview for assessing suicidal ideation, min value=0, max value = 38. Higher score = worse outcome.

SECONDARY OUTCOMES:
Change in Scale for Suicidal Ideation Change | Change from baseline, to end of TBS treatment course (4 weeks), and at 1 month follow up
  A semi-structured interview for assessing suicidal ideation, min value=0, max value = 38. Higher score = worse outcome.
Change in Columbia - Suicide Severity Rating Scale Change | Change from baseline, to end of TBS treatment course (4 weeks), and at 1 month follow up
  An interviewer-rated suicide risk assessment tool. Min value = 0, Max value = N/A. Higher score = worse outcome
17-item Hamilton Rating Scale for Depression (HRSD-17) Change | Baseline, after TBS treatment course (4 weeks), and at 1 month follow up
  A rating scale for measuring severity of depressive symptoms. Min value = 0 Max value = 52. Higher score = worse outcome
Visual Analogue Scale for Opioid Cravings Change | Baseline, after TBS treatment course (4 weeks), and at 1 month follow up
  A rating scale for subjective cravings to use opioids. Min value = 0 Max value = 100. Higher score = worse outcome.
Timeline Followback Change | Baseline, after TBS treatment course (4 weeks), and at 1 month follow up
  Self-reported substance use over a designated period of time. Min value = 0 Max value = N/A. Higher score = worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Voineskos, MD, PhD, Principal Investigator — Clinician Scientist, Psychiatrist
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tang VM, Le Foll B, Daskalakis ZJ, Wang AL, Buckley L, Blumberger DM, Voineskos D. Repetitive transcranial magnetic stimulation for the treatment of suicidality in opioid use disorder: a pilot feasibility randomized controlled trial. Eur Psychiatry. 2025 Mar 5;68(1):e63. doi: 10.1192/j.eurpsy.2025.28. PMID 40040511